CLINICAL TRIAL: NCT02371629
Title: A Randomized, Double-blind, Parallel Group, 26-week Study Evaluating the Efficacy, Safety and Tolerability of NVA237 Given Once or Twice Daily, in Patients With Moderate and Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study of the Efficacy and Safety of NVA237 in Patients With Moderate to Severe COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A2320
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Anticholinergic; Antimuscarinic; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; COPD; LAMA; Lung Disease; Lung Diseases, Obstructive; Lung Function; Muscarinic receptor antagonist; Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive; Respiratory Tract Diseases | interventions — Glycopyrrolate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 Twice daily (Experimental): Patients randomized to this arm received an NVA237 22 μg capsule in the morning and evening for 26 weeks. All participants received salbutamol as rescue medicine.
  Interventions: Drug: NVA237; Drug: Salbutamol
- NVA237 Once daily (Experimental): Patients randomized to this arm received an NVA237 44 μg capsule in the morning and a placebo capsule in the evening for 26 weeks. All participants received salbutamol as rescue medicine.
  Interventions: Drug: NVA237; Drug: Placebo; Drug: Salbutamol

INTERVENTIONS:
Drug: NVA237 — NVA237 capsules for inhalation, delivered via a Single Dose Dry Powder Inhaler (SDDPI) called Concept1
  Other Names: glycopyrronioum bromide
Drug: Placebo — Placebo to NVA237
  Arms: NVA237 Once daily
Drug: Salbutamol — All patients received salbutamol (100 μg) as only rescue medication

SUMMARY:
This study is a post-authorization commitment to the European Medicines Agency (EMA). The study serves to determine whether the treatment of patients with stable, symptomatic Chronic Obstructive Pulmonary Disease (COPD) with the investigational drug NVA237 is efficient and safe. The efficacy and safety of the drug was tested for twice daily dosing against once daily dosing.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Male and female adults aged ≥40 years
* Patients with stable COPD according to the current GOLD strategy (GOLD 2014)
* Current or ex-smokers who have a smoking history of at least 10 pack years- an ex-smoker may be defined as a subject who has not smoked for ≥ 6 months at screening
* mMRC grade of at least 2 at Visit 101
* Patients with airflow limitation indicated by a post-bronchodilator FEV1 ≥ 30 % and < 80 % of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70 at Visit 101.

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test; Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment
* Patients with Type I or uncontrolled Type II diabetes; Patients with a history of long QT syndrome or whose QTc measured at run-in (Fridericia method) is prolonged (>450 ms for males and >460 for females) and confirmed by a central assessor
* Patients requiring long term oxygen therapy prescribed for >12 h per day; Patients with any history of asthma.

Ages: 41 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- Belgium (2):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Jambes, Namur
- Bulgaria (17):
  - Novartis Investigative Site, Sevlievo, Gabrovo
  - Novartis Investigative Site, Sofia, Sofia-Grad
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Kozloduy
  - Novartis Investigative Site, Lom
  - Novartis Investigative Site, Lovech
  - Novartis Investigative Site, Montana
  - Novartis Investigative Site, Razgrad
  - Novartis Investigative Site, Roman
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Silistra
  - Novartis Investigative Site, Sliven
  - Novartis Investigative Site, Smolyan
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Troyan Municipality
  - Novartis Investigative Site, Veliko Tarnovo
  - Novartis Investigative Site, Vidin
- Novartis Investigative Site, Turku, Finland
- Germany (11):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Großhansdorf, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Wiesbaden
- Hungary (7):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Farkasgyepű
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Sopron
  - Novartis Investigative Site, Szarvas
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Rehovot, Israel
- Poland (10):
  - Novartis Investigative Site, Tarnów, Lesser Poland Voivodeship
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Lodz, Lódzkie
  - Novartis Investigative Site, Chorzów, Silesian Voivodeship
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Wilkowice
- Romania (7):
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Tg Mures, Mureș County
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (11):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yaroslavl
- Sweden (5):
  - Novartis Investigative Site, Malmo, Skåne County
  - Novartis Investigative Site, Lidingo, Södermanland County
  - Novartis Investigative Site, Gothenburg, Västra Götaland County
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Linköping, Östergötland County

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1020 patients were screened for participation in this study; 776 were randomized.
Period: Overall Study
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Started | 388 | 388
Completed | 362 | 363
Not Completed | 26 | 25
Not completed — Patient decision | 14 | 10
Not completed — Adverse Event | 8 | 8
Not completed — Physician Decision | 2 | 3
Not completed — Death | 1 | 1
Not completed — Noncompliance with study treatment | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily | Total
Number analyzed (Participants) | 388 | 388 | 776
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.71) | 63.6 (7.66) | 63.4 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 111 | 233
  Male | 266 | 277 | 543

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: Spirometry testing was performed in accordance with American Thoracic Society standards. Trough FEV1 defined as the mean of two measurements at 23 hours 15 minutes and 23 hour 45 minutes post dosing. Baseline FEV1 was defined as the average of the -45 minutes and -15 minutes FEV1 values taken on Day 1. An analysis-of-covariance (ANCOVA) for repeated measurements, also known as mixed model for repeated measures (MMRM), was performed for the change from baseline of trough FEV1 at Week 12. The model included treatment, COPD severity, baseline smoking status, baseline ICS use, region, and visit (Day 1, and Weeks 12 and 26) as factors and baseline FEV1 as a covariate.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and week 12 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 358 | 360
Liters | 0.092 (0.0126) | 0.059 (0.0125)
Statistical Analysis 1: Comparison: NVA237 Twice Daily vs NVA237 Once Daily; Test type: Superiority or Other; p = 0.051, Mixed model for repeated measure (MMRM); Mean Difference (Net) = 0.033, 95% CI 2-sided [0.000 to 0.066], Standard Error of Mean 0.0169

2. Secondary Outcome: Change From Baseline in Area Under The Curve (AUC) for Forced Expiratory Volume in One Second (FEV1) for Different Time Spans Post Dosing at Week 12
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) is assessed for different time spans (0-12h, 0-24h, 12-24h) within the overall serial measurement post dosing at week 12 of treatment. Baseline FEV1 was defined as the average of the -45 minutes and -15 minutes FEV1 values taken on Day 1.
Time Frame: Baseline, 0-12 hour, 0-24 hour , 12-24 hour post dose at Week 12
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at baseline and week 12 in different time spans were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 373 | 373
Liters
  AUC (0-12 hour) | 0.136 (0.0119) | 0.106 (0.0118)
  AUC (0-24 hour) | 0.085 (0.0121) | 0.043 (0.0120)
  AUC (12-24 hour): number analyzed (Participants) | 371 | 371
  AUC (12-24 hour) | 0.035 (0.0125) | -0.019 (0.0124)

3. Secondary Outcome: Change From Baseline in Area Under The Curve (AUC 0-12 Hour) for Forced Expiratory Volume in One Second (FEV1) Post Dosing at Day 1
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) is assessed for 0-12 hour, post dosing at Day 1 of treatment. Baseline FEV1 was defined as the average of the -45 minutes and -15 minutes FEV1 values taken on Day 1.
Time Frame: Baseline, 0-12 hour post dose at Day 1
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and Day 1 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 387 | 387
Liters | 0.143 (0.0089) | 0.139 (0.0087)

4. Secondary Outcome: Change From Baseline in Area Under The Curve (AUC) for Forced Expiratory Volume in One Second (FEV1) for Different Time Spans Post Dosing at Week 26
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) is assessed for different time spans (0-12h, 0-24h, 12-24h) within the overall serial measurement post dosing at week 26 of treatment. Baseline FEV1 was defined as the average of the -45 minutes and -15 minutes FEV1 values taken on Day 1.
Time Frame: Baseline, 0-12 hour, 0-24 hour , 12-24 hour post dose at Week 26
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and week 26 in different time spans were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 360 | 364
Liters
  AUC (0-12 hour): number analyzed (Participants) | 360 | 363
  AUC (0-12 hour) | 0.123 (0.0121) | 0.091 (0.0120)
  AUC (0-24 hour) | 0.076 (0.0122) | 0.030 (0.0121)
  AUC (12-24 hour): number analyzed (Participants) | 357 | 361
  AUC (12-24 hour) | 0.032 (0.0127) | -0.028 (0.0126)

5. Secondary Outcome: Change From Baseline in Total St. George's Respiratory Questionnaire (SGRQ) Score at Week 12 and Week 26
Description: The health status, as reported by the patients, is assessed using the St. George's Respiratory Questionnaire (SGRQ). The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD:
  * Part I covers "Symptoms" and is concerned with respiratory symptoms, their frequency and severity
  * Part II covers "Activity" and is concerned with activities that caused or are limited by breathlessness
  * Part II is also concerned with "Impacts", which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease.
  A score was calculated for each of these three subscales and the total score was calculated. In each case, the lowest possible value was 0 and the highest 100. Higher values corresponded to greater impairment of health status.
Time Frame: Baseline, 12 Weeks, 26 Weeks
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and post-baseline time points were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
score on a scale
  Change from Baseline to WK 12: number analyzed (Participants) | 369 | 369
  Change from Baseline to WK 12 | -5.320 (0.6000) | -3.563 (0.5987)
  Change from Baseline to WK 26: number analyzed (Participants) | 357 | 359
  Change from Baseline to WK 26 | -6.587 (0.6543) | -4.644 (0.6527)

6. Secondary Outcome: Percentage of Patients With a Clinically Significant Improvement in St George Respiratory Questionnaire at Week 12 and Week 26
Description: The health status, as reported by the patients, is assessed using the St. George's Respiratory Questionnaire (SGRQ).
  The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD:
  * Part I covers "Symptoms" and is concerned with respiratory symptoms, their frequency and severity
  * Part II covers "Activity" and is concerned with activities that caused or are limited by breathlessness
  * Part II is also concerned with "Impacts", which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease.
  A score was calculated for each of these three subscales and the total score was calculated. In each case, the lowest possible value was 0 and the highest 100.
  A clinically significant improvement is defined as ≥ 4 unit improvement from baseline score (a decrease of ≥ 4).
Time Frame: Baseline, 12 Weeks, 26 Weeks
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. n= the number of patients with a SGRQ total score at both baseline and indicated post-baseline time point
Measure: Number; unit: percentage of patients
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
percentage of patients
  Change from Baseline to WK 12: number analyzed (Participants) | 369 | 369
  Change from Baseline to WK 12 | 54.5 | 46.9
  Change from Baseline to WK 26: number analyzed (Participants) | 357 | 359
  Change from Baseline to WK 26 | 59.4 | 49.6

7. Secondary Outcome: Change From Baseline in Transitional Dyspnea Index (TDI) Focal Score at Week 12 and Week 26
Description: Breathlessness at Week 12 and Week 26 is measured using the Transition Dyspnea Index (TDI). On day 1, breathlessness is assessed by the Baseline Dyspnea Index (BDI). Baseline Dyspnea Index (BDI)/Transition Dyspnea Index (TDI) focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort and captures changes from baseline. BDI was measured at day 1 prior to the first dose with domain scores ranging from 0=very severe to 4=no impairment and a total score ranging from 0 to 12(best). TDI captures changes from baseline. Each domain is scored from -3=major deterioration to 3=major improvement to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score.
Time Frame: Baseline, 12 Weeks, 26 Weeks
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and post-baseline time points were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
score on a scale
  Change from Baseline to WK 12: number analyzed (Participants) | 360 | 356
  Change from Baseline to WK 12 | 1.346 (0.1430) | 0.849 (0.1433)
  Change from Baseline to WK 26: number analyzed (Participants) | 347 | 348
  Change from Baseline to WK 26 | 1.523 (0.1539) | 1.170 (0.1534)

8. Secondary Outcome: Percentage of Patients With a Clinically Important Improvement on Transitional Dyspnea Index (TDI) Focal Score at Week 12 and Week 26
Description: Breathlessness at Week 12 and Week 26 is measured using the Transition Dyspnea Index (TDI). On day 1, breathlessness is assessed by the Baseline Dyspnea Index (BDI). Baseline Dyspnea Index (BDI)/Transition Dyspnea Index (TDI) focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort and captures changes from baseline. BDI was measured at day 1 prior to the first dose with domain scores ranging from 0=very severe to 4=no impairment and a total score ranging from 0 to 12(best). TDI captures changes from baseline. Each domain is scored from -3=major deterioration to 3=major improvement to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score.
  Clinically important improvement indicates ≥ 1 unit in the TDI focal score at Weeks 12 and 26 in comparison to BDI focal score (an increase of ≥ 1).
Time Frame: Baseline, 12 Weeks, 26 Weeks
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. n= the number of patients with a TDI focal score
Measure: Number; unit: Percentage of patients
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
Percentage of patients
  Change from Baseline to WK 12: number analyzed (Participants) | 360 | 356
  Change from Baseline to WK 12 | 56.9 | 52.0
  Change from Baseline to WK 26: number analyzed (Participants) | 347 | 348
  Change from Baseline to WK 26 | 61.1 | 54.6

9. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 1 and Week 26
Description: Spirometry testing was performed in accordance with American Thoracic Society standards. Trough FEV1 defined as the mean of two measurements at 23 hours 15 minutes and 23 hour 45 minutes post dosing. Baseline FEV1 was defined as the average of the -45 minutes and -15 minutes FEV1 values taken on Day 1. An analysis-of-covariance (ANCOVA) for repeated measurements, also known as mixed model for repeated measures (MMRM), was performed for the change from baseline of trough FEV1. The model included treatment, COPD severity, baseline smoking status, baseline ICS use, region, and visit (Day 1, and Weeks 12 and 26) as factors and baseline FEV1 as a covariate.
Time Frame: Baseline, Day 1, Week 26
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
Liters
  Change from baseline to Day 1: number analyzed (Participants) | 381 | 381
  Change from baseline to Day 1 | 0.119 (0.0099) | 0.070 (0.0097)
  Change from baseline to Week 26: number analyzed (Participants) | 341 | 349
  Change from baseline to Week 26 | 0.104 (0.0129) | 0.056 (0.0128)

10. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Individual Timepoints at Week 26
Description: Mixed model for repeated measures was used to analyze change from baseline in FVC. Baseline FVC is defined as the average of the -45 min and -15 min FVC values taken on Day 1 prior to first dose.
Time Frame: Baseline, Week 26 (Day 183-184)
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following intent-to-treat principle, patients in FAS were analyzed according to the treatment to which they were randomized. n = number of patients included in respective analysis (i.e. who had a FVC at this time point on at least one visit).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
Liters
  Day 183/-45 min:: number analyzed (Participants) | 334 | 342
  Day 183/-45 min: | 0.079 (0.0195) | 0.025 (0.0192)
  Day 183/-15 min:: number analyzed (Participants) | 340 | 345
  Day 183/-15 min: | 0.102 (0.0193) | 0.029 (0.0191)
  Day 183/5 min:: number analyzed (Participants) | 335 | 337
  Day 183/5 min: | 0.159 (0.0194) | 0.085 (0.0194)
  Day 183/15 min:: number analyzed (Participants) | 333 | 334
  Day 183/15 min: | 0.177 (0.0195) | 0.132 (0.0195)
  Day 183/30 min:: number analyzed (Participants) | 344 | 346
  Day 183/30 min: | 0.194 (0.0192) | 0.144 (0.0191)
  Day 183/1 h:: number analyzed (Participants) | 335 | 343
  Day 183/1 h: | 0.190 (0.0194) | 0.154 (0.0192)
  Day 183/2 h: number analyzed (Participants) | 340 | 345
  Day 183/2 h | 0.229 (0.0193) | 0.200 (0.0191)
  Day 183/3 h:: number analyzed (Participants) | 327 | 344
  Day 183/3 h: | 0.229 (0.0197) | 0.186 (0.0192)
  Day 183/4 h:: number analyzed (Participants) | 335 | 347
  Day 183/4 h: | 0.216 (0.0194) | 0.169 (0.0191)
  Day 183/6 h: number analyzed (Participants) | 330 | 347
  Day 183/6 h | 0.146 (0.0196) | 0.116 (0.0191)
  Day 183/8 h: number analyzed (Participants) | 331 | 341
  Day 183/8 h | 0.137 (0.0195) | 0.085 (0.0193)
  Day 183/10 h: number analyzed (Participants) | 323 | 345
  Day 183/10 h | 0.071 (0.0198) | 0.039 (0.0191)
  Day 183/12 h: number analyzed (Participants) | 318 | 331
  Day 183/12 h | 0.041 (0.0200) | 0.026 (0.0196)
  Day 183/13 h: number analyzed (Participants) | 320 | 326
  Day 183/13 h | 0.096 (0.0199) | 0.004 (0.0197)
  Day 184/16 h: number analyzed (Participants) | 295 | 298
  Day 184/16 h | -0.014 (0.0207) | -0.081 (0.0206)
  Day 184/22 h: number analyzed (Participants) | 323 | 333
  Day 184/22 h | -0.036 (0.0198) | -0.076 (0.0195)
  Day 184/23 h 15 min: number analyzed (Participants) | 314 | 336
  Day 184/23 h 15 min | 0.075 (0.0201) | 0.031 (0.0194)
  Day 184/23 h 45 min: number analyzed (Participants) | 325 | 329
  Day 184/23 h 45 min | 0.129 (0.0197) | 0.077 (0.0196)

11. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC) at Individual Timepoints at Week 26
Description: Mixed model for repeated measures was used to analyze change from baseline in IC.
Time Frame: Baseline, Week 26 (Day 183-184)
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following intent-to-treat principle, patients in FAS were analyzed according to the treatment to which they were randomized. n = number of patients included in respective analysis (i.e. who had a IC at this timepoint on at least one visit).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
Liters
  Day 183/-20 min: number analyzed (Participants) | 225 | 224
  Day 183/-20 min | 0.094 (0.0221) | 0.054 (0.0221)
  Day 183/25 min: number analyzed (Participants) | 220 | 237
  Day 183/25 min | 0.181 (0.0224) | 0.173 (0.0215)
  Day 183/1 h 55 min: number analyzed (Participants) | 222 | 232
  Day 183/1 h 55 min | 0.193 (0.0223) | 0.171 (0.0218)
  Day 183/3 h 55 min: number analyzed (Participants) | 215 | 225
  Day 183/3 h 55 min | 0.163 (0.0226) | 0.159 (0.0221)
  Day 183/7 h 55 min: number analyzed (Participants) | 213 | 223
  Day 183/7 h 55 min | 0.108 (0.0228) | 0.110 (0.0222)
  Day 183/11 h 55 min: number analyzed (Participants) | 210 | 231
  Day 183/11 h 55 min | 0.042 (0.0229) | 0.030 (0.0218)
  Day 184/23 h 40 min: number analyzed (Participants) | 203 | 221
  Day 184/23 h 40 min | 0.045 (0.0233) | 0.062 (0.0224)

12. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at Individual Timepoints at Week 26
Description: Mixed model for repeated measures was used to analyze change from baseline in FEV1. Baseline FEV1 is defined as the average of the -45 min and -15 min FEV1 values taken on Day 1 prior to first dose.
Time Frame: Baseline, Week 26 (Day 183-184)
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following intent-to-treat principle, patients in FAS were analyzed according to the treatment to which they were randomized. n = number of patients included in respective analysis (i.e. who had a FEV1 at this timepoint on at least one visit).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
Liters
  Day 183/-45 min: number analyzed (Participants) | 334 | 342
  Day 183/-45 min | 0.058 (0.0120) | 0.012 (0.0119)
  Day 183/-15 min: number analyzed (Participants) | 340 | 345
  Day 183/-15 min | 0.086 (0.0119) | 0.034 (0.0118)
  Day 183/5 min: number analyzed (Participants) | 335 | 337
  Day 183/5 min | 0.111 (0.0120) | 0.070 (0.0119)
  Day 183/15 min: number analyzed (Participants) | 333 | 334
  Day 183/15 min | 0.145 (0.0120) | 0.106 (0.0120)
  Day 183/30 min: number analyzed (Participants) | 344 | 346
  Day 183/30 min | 0.155 (0.0118) | 0.122 (0.0118)
  Day 183/1 h: number analyzed (Participants) | 335 | 343
  Day 183/1 h | 0.158 (0.0120) | 0.132 (0.0118)
  Day 183/2 h: number analyzed (Participants) | 340 | 345
  Day 183/2 h | 0.194 (0.0119) | 0.163 (0.0118)
  Day 183/3 h: number analyzed (Participants) | 327 | 344
  Day 183/3 h | 0.179 (0.0121) | 0.154 (0.0118)
  Day 183/4 h: number analyzed (Participants) | 335 | 347
  Day 183/4 h | 0.166 (0.0120) | 0.132 (0.0118)
  Day 183/6 h: number analyzed (Participants) | 330 | 347
  Day 183/6 h | 0.110 (0.0121) | 0.080 (0.0118)
  Day 183/8 h: number analyzed (Participants) | 331 | 341
  Day 183/8 h | 0.118 (0.0121) | 0.064 (0.0119)
  Day 183/10 h: number analyzed (Participants) | 323 | 345
  Day 183/10 h | 0.067 (0.0122) | 0.038 (0.0118)
  Day 183/12 h: number analyzed (Participants) | 318 | 331
  Day 183/12 h | 0.056 (0.0123) | 0.024 (0.0121)
  Day 183/13 h: number analyzed (Participants) | 320 | 326
  Day 183/13 h | 0.093 (0.0123) | 0.000 (0.0121)
  Day 184/16 h: number analyzed (Participants) | 295 | 298
  Day 184/16 h | -0.001 (0.0128) | -0.063 (0.0127)
  Day 184/22 h: number analyzed (Participants) | 323 | 333
  Day 184/22 h | -0.012 (0.0122) | -0.043 (0.0120)
  Day 184/23 h 15 min: number analyzed (Participants) | 314 | 336
  Day 184/23 h 15 min | 0.076 (0.0124) | 0.032 (0.0120)
  Day 184/23 h 45 min: number analyzed (Participants) | 325 | 329
  Day 184/23 h 45 min | 0.122 (0.0122) | 0.067 (0.0121)

13. Secondary Outcome: Change From Baseline in the Percentage of Days With no Rescue Medication Use Over the 26 Weeks
Description: Patients report the number of puffs of rescue medication (salbutamol / albuterol) using an electronic diary. change from baseline in percentage of days without rescue medication usage over 26 weeks was analyzed.
Time Frame: Baseline, 26 Weeks
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and week 26 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 383 | 377
percentage of days | 16.574 (2.3519) | 15.363 (2.3927)

14. Secondary Outcome: Change From Baseline in Mean Daily COPD Symptom Score at Week 26
Description: Patients reported symptoms by using an electronic diary. The mean daily total symptom score, the mean morning symptom score and the mean evening symptom score were calculated for each patient over 26 weeks. Each symptom measured in a numeric rating scale of 0-10; 0 indicates no symptom and 10 indicates severe symptom. 0 is no waking due to symptoms, 1 woke up once, 2 woke up more than once due to symptoms ; 10 was the worst score.The daily score for an individual symptom score was the worst of the morning and evening scores on a particular day. If either the morning or evening score was missing for a symptom then the non-missing value was taken as the worst. A negative change indicates improvement. Only the scores for the 6 COPD symptoms (respiratory symptoms, cough, wheeze, production of sputum, sputum color, and breathlessness) were used to derive the total symptom score
Time Frame: Baseline, 26 Weeks
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients in the FAS were analyzed according to the treatment to which they were randomized. Patients with evaluable data at both baseline and week 26 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 383 | 377
score on a scale
  Change in mean daily | -1.336 (0.1141) | -1.107 (0.1160)
  Change in mean morning: number analyzed (Participants) | 374 | 374
  Change in mean morning | -1.032 (0.1304) | -0.828 (0.1318)
  Change in mean evening: number analyzed (Participants) | 372 | 375
  Change in mean evening | -1.205 (0.1141) | -1.056 (0.1152)

15. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death
Description: This endpoint reports patients affected by any adverse events (AE), serious adverse events (SAE) and death. Only treatment emergent AE, SAE, deaths are reported for this endpoint.
Time Frame: 26 Weeks
Population: The Safety Set (SAF) included all patients who received at least one dose of study drug whether or not they were randomized. Patients were analyzed according to the treatment they received. If patients switched treatment during the study, they were to be analyzed according to the treatment to which they were randomized.
Measure: Number; unit: Count of Participants
Arm/Group | NVA237 Twice Daily | NVA237 Once Daily
Number analyzed (Participants) | 388 | 388
Count of Participants
  Patients with at least one AE | 203 | 224
  Patients with at least one SAE | 33 | 30
  Death | 1 | 1

ADVERSE EVENTS:
Groups:
- NVA237 22 mcg b.i.d.: NVA237 22 mcg b.i.d.
- NVA237 44 mcg o.d.: NVA237 44 mcg o.d.
Arm/Group | NVA237 22 mcg b.i.d. | NVA237 44 mcg o.d.
All-Cause Mortality (participants affected / at risk) | 1/388 | 2/388
Serious Adverse Events (participants affected / at risk) | 33/388 | 30/388
Other Adverse Events (participants affected / at risk) | 126/388 | 152/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 22 mcg b.i.d. (N=388) | NVA237 44 mcg o.d. (N=388)
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4
Sepsis (Infections and infestations) | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Pseudoradicular syndrome (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 15
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Brachiocephalic artery stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 22 mcg b.i.d. (N=388) | NVA237 44 mcg o.d. (N=388)
Bronchitis (Infections and infestations) | 10 | 3
Nasopharyngitis (Infections and infestations) | 37 | 54
Headache (Nervous system disorders) | 4 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 74 | 99
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Hypertension (Vascular disorders) | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.